CLINICAL TRIAL: NCT06536192
Title: Improving Gynecological Examination Skills in Midwifery Students: a Training Study Using Models
Brief Title: Improving Gynecological Examination Skills with the Use of a Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ayse Cuvadar, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E-77192459-050.99-338662
Record Dates: First submitted 2024-07-22; First posted 2024-08-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Nursing; Training Group, Sensitivity; Gynecologic Disease
Keywords: Midwife, student, gynecological examination, model
MeSH Terms: conditions — Hypersensitivity; Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Model) group (Experimental): 1. Process: Theoretical knowledge will be given to students, and then different types of gynecological examinations will be explained practically on a model in the laboratory environment.
  2. Process: The learner guide will be filled out.
  3. Process: After 15 days, students will be taken back to the laboratory environment to fill out the learner guide again. In addition, Self-Confidence Scale (SCS) and Student Satisfaction and Self-Confidence in Learning Scale (SSSLS) will be filled out for the last exam.
  Interventions: Other: Model group
- Control group (No Intervention): 1. Procedure: The stages of gynecological examination evaluation for students, its purpose, the process of preparing the patient and evaluating them will be provided with theoretical knowledge.
  2. Procedure: Pre-tests will be administered.
  3. Procedure: Two weeks later, Self-Confidence Scale (SCS); Learner's Guide (LG) and (Student Satisfaction and Self-Confidence in Learning Scale) SSSCLS will be filled out for the final test.

INTERVENTIONS:
Other: Model group — 1. Process: Theoretical knowledge will be given to students, and then different types of gynecological examinations will be explained practically on a model in the laboratory environment.
  2. Process: The learner guide will be filled out.
  3. Process: After 15 days, students will be taken back to the laboratory environment to fill out the learner guide again. In addition, SCS and SSSLS will be filled out for the last exam.
  Arms: Intervention (Model) group

SUMMARY:
Vaginal, abdominal, and breast examinations are among the essential gynecological examination skills for midwifery students and are crucial steps that need to be learned. However, due to the privacy of genital areas, there are some debates regarding the teaching of these skills. Low-fidelity mannequins and models are particularly effective and cost-efficient in acquiring basic psychomotor skills. Thus, midwifery students can gain clinical experience, make mistakes in a safe environment, and enhance their skills. The sample of this study consists of 64 midwifery students (experimental=32, control=32) using a pre-test, post-test design with an observational randomized controlled trial. Data collection instruments include a Personal Information Form (PIF), Learner's Guide (LG), Self-Confidence Scale (SCS), and Self-Confidence in Learning Scale (SSSCLS. In the experimental group, after providing theoretical knowledge, students will receive practical training on a gynecological examination model, including bimanual examination, vaginal examination with a speculum, pap smear for cervical screening, and pelvic palpation. Each student will then perform the examination individually, with approximately 15 minutes allocated per student. Two weeks later, the same students will be asked to perform all examination steps again. During the examinations, the researcher will mark complete and incomplete procedures in the learner's guide, and any deficiencies will be explained to the students for completion. The CS and SSSLS will be administered for the post-test. In the control group, after theoretical knowledge is provided, students will be shown visual and video demonstrations of the steps of a gynecological examination. The PIF and SCS will be administered for the pre-test, and two weeks later, students will be asked to perform the examination steps in a laboratory setting, followed by the post-test.

DETAILED DESCRIPTION:
Gynecological examination is an important step for women's health. Early diagnosis, treatment, intervention, and follow-up are the foundation of a healthy life. Midwives play an important role in maintaining women's health, especially in conducting detailed gynecological and obstetric evaluations. They should receive quality theoretical education and improve their practices. Practical training is important in learning, especially in the health field where models and simulation applications play a significant role in clinical practices. Therefore, clinical examination skills are sometimes taught to students using different materials, making it easier for students to learn medical knowledge and reducing the time spent on education. The aim of this planned study is to improve midwifery students' gynecological examination skills with model support.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd or 4th year midwifery student at Karabük University Faculty of Health Sciences

  * Being between the ages of 18-25
  * Voluntarily agreeing to participate in the study
  * Being a citizen of the Republic of Turkey

Exclusion Criteria:

* Leave whenever you want without working.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Improving gynecological examination skills with the use of a model | Groups of 5 people receive 15 minutes of laboratory training and 15 days later, practice in the laboratory.
  Gynecologic Disease

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Karabük University, Karabük, Karabük Province
  - Ayşe Çuvadar, Karabük, Turkey

IPD SHARING:
Plan to Share IPD: No